CLINICAL TRIAL: NCT03303794
Title: Comparative Feasibility and Efficacy of a Five Compartment Technique Using 0.25% Bupivacaine vs a Mixture of 0.25% Bupivacaine and 1.3 % Liposomal Bupivacaine in Patients Undergoing Tka; a Single Blinded Randomized Controlled Study
Brief Title: 0.25% Bupivacaine Versus a Mixture of 0.25% Bupivacaine and 1.3 % Liposomal Bupivacaine in Patients Undergoing Tka
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim Analysis showed no significance
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Singh Nair, Investigator, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-7893
Record Dates: First submitted 2017-09-26; First posted 2017-10-06 (Actual); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Anesthesia
Keywords: Total Knee arthroplasty; bupivacaine; anesthesia
MeSH Terms: interventions — Bupivacaine; Liposomes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivicaine (Active Comparator): 0.25% bupivacaine in patients undergoing total knee arthroplasty
  Interventions: Drug: 0.25% bupivacaine
- Bupivicaine + Exparel (Experimental): 0.25% bupivacaine and 1.3 % liposomal Bupivacaine in patients undergoing total knee arthroplasty
  Interventions: Drug: Exparel; Drug: 0.25% bupivacaine

INTERVENTIONS:
Drug: Exparel — 1.3 % liposomal Bupivacaine in patients undergoing total knee arthroplasty
  Arms: Bupivicaine + Exparel
Drug: 0.25% bupivacaine — 0.25% bupivacaine in patients undergoing total knee arthroplasty
  Other Names: liposomal

SUMMARY:
Total knee and hip replacements are some of the most common orthopedic procedures that require aggressive postoperative pain management. This management helps us to improve clinical outcomes such as participation in early physical therapy, hospital discharge, and patient satisfaction. Based on the recent anatomical evidence and the investigator's knowledge of the complexity of the knee joint innervation the investigator proposes a new regional anesthesia technique that provides a complete sensory blockade and better analgesia while preserving the quadriceps strength and avoiding the potential for foot drop caused by inadvertent blockade of the common peroneal nerve.

DETAILED DESCRIPTION:
This is an assessor-blinded randomized controlled trial evaluating the efficacy of liposomal bupivacaine (Exparel) in patients undergoing Total Knee Arthroplasty. The primary outcome of this study is the proportion of patients "fit to discharge" on postoperative day one. Recently, liposomal bupivacaine (LB) (Exparel) was introduced into clinical practice, using a lipid-based depot (DepoFoam) technology for sustained release of bupivacaine. LB (Exparel) uses this technology to extend the delivery of bupivacaine, a local anesthetic that has been used in clinical practice for decades for peripheral nerve block, spinal, and epidural analgesia and anesthesia. This formulation prolongs the duration of analgesia of bupivacaine for up to 72 hours with a single injection. The study was designed to compare two of our current standard therapies:

1. Adductor Canal Block + Tissue Infiltration (lateral, medial and femoral compartment + posterior capsule tissue infiltration using 0.25% bupivacaine; and
2. Adductor Canal Block + Tissue Infiltration (lateral, medial and femoral compartment + posterior capsule tissue infiltration) using 1:1 mixture of 1.3% LB (Exparel) + 0.5% bupivacaine HCl mixture.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing unilateral total knee replacement due to OA or rheumatoid arthritis
* Ages 40- 80 years old
* American Society of Anesthesiologists class I-III

Exclusion Criteria:

* Refusal or absolute medical contraindication to peripheral nerve block
* refusal or absolute medical contraindication to spinal anesthesia
* conversion of spinal anesthesia to general anesthesia is obtained
* inability to cooperate
* allergy to any drug used in this study
* daily intake of opioids (tramadol, morphine, oxycodone, methadone, fentanyl)
* alcohol dependence or use of any illegal drugs within the last month
* inability to perform the mobilization test and timed up and go (TUG) test pre-operatively

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boleslav Kosharskyy, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Hutchinson Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
All study data will be collected and entered into the computer database. Each subject will be assigned to a random number code and the key linking the code and the subject identifier will be stored in a locked cabinet. The computer database will be password protected and will be kept on the Montefiore drive. The research manager is responsible for auditing the consistency of the data transcribed from the paper case report form to the computer. A protocol violation log will be maintained and all protocol violations will be reported to the Institutional Review Board and Data Safety Monitoring Board. The planned interim analysis (half way through the recruitment) will be mainly focused on the adverse events, rather than the efficacy of the procedure.

REFERENCES:
- [Background] Johnson RL, Kopp SL, Hebl JR, Erwin PJ, Mantilla CB. Falls and major orthopaedic surgery with peripheral nerve blockade: a systematic review and meta-analysis. Br J Anaesth. 2013 Apr;110(4):518-28. doi: 10.1093/bja/aet013. Epub 2013 Feb 24. PMID 23440367
- [Background] Hebl JR, Dilger JA, Byer DE, Kopp SL, Stevens SR, Pagnano MW, Hanssen AD, Horlocker TT. A pre-emptive multimodal pathway featuring peripheral nerve block improves perioperative outcomes after major orthopedic surgery. Reg Anesth Pain Med. 2008 Nov-Dec;33(6):510-7. PMID 19258965
- [Background] Hebl JR, Kopp SL, Ali MH, Horlocker TT, Dilger JA, Lennon RL, Williams BA, Hanssen AD, Pagnano MW. A comprehensive anesthesia protocol that emphasizes peripheral nerve blockade for total knee and total hip arthroplasty. J Bone Joint Surg Am. 2005;87 Suppl 2:63-70. doi: 10.2106/JBJS.E.00491. No abstract available. PMID 16326725
- [Background] Ilfeld BM, Le LT, Meyer RS, Mariano ER, Vandenborne K, Duncan PW, Sessler DI, Enneking FK, Shuster JJ, Theriaque DW, Berry LF, Spadoni EH, Gearen PF. Ambulatory continuous femoral nerve blocks decrease time to discharge readiness after tricompartment total knee arthroplasty: a randomized, triple-masked, placebo-controlled study. Anesthesiology. 2008 Apr;108(4):703-13. doi: 10.1097/ALN.0b013e318167af46. PMID 18362603
- [Background] Feibel RJ, Dervin GF, Kim PR, Beaule PE. Major complications associated with femoral nerve catheters for knee arthroplasty: a word of caution. J Arthroplasty. 2009 Sep;24(6 Suppl):132-7. doi: 10.1016/j.arth.2009.04.008. Epub 2009 Jun 24. PMID 19553071
- [Background] Ilfeld BM, Ball ST, Gearen PF, Le LT, Mariano ER, Vandenborne K, Duncan PW, Sessler DI, Enneking FK, Shuster JJ, Theriaque DW, Meyer RS. Ambulatory continuous posterior lumbar plexus nerve blocks after hip arthroplasty: a dual-center, randomized, triple-masked, placebo-controlled trial. Anesthesiology. 2008 Sep;109(3):491-501. doi: 10.1097/ALN.0b013e318182a4a3. PMID 18719448
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Kandasami M, Kinninmonth AW, Sarungi M, Baines J, Scott NB. Femoral nerve block for total knee replacement - a word of caution. Knee. 2009 Mar;16(2):98-100. doi: 10.1016/j.knee.2008.10.007. Epub 2008 Nov 28. PMID 19046884
- [Background] Klein SM, Nielsen KC, Greengrass RA, Warner DS, Martin A, Steele SM. Ambulatory discharge after long-acting peripheral nerve blockade: 2382 blocks with ropivacaine. Anesth Analg. 2002 Jan;94(1):65-70, table of contents. doi: 10.1097/00000539-200201000-00012. PMID 11772802
- [Background] Muraskin SI, Conrad B, Zheng N, Morey TE, Enneking FK. Falls associated with lower-extremity-nerve blocks: a pilot investigation of mechanisms. Reg Anesth Pain Med. 2007 Jan-Feb;32(1):67-72. doi: 10.1016/j.rapm.2006.08.013. PMID 17196495
- [Background] Sharma S, Iorio R, Specht LM, Davies-Lepie S, Healy WL. Complications of femoral nerve block for total knee arthroplasty. Clin Orthop Relat Res. 2010 Jan;468(1):135-40. doi: 10.1007/s11999-009-1025-1. Epub 2009 Aug 13. PMID 19680735
- [Background] Williams BA, Kentor ML, Bottegal MT. The incidence of falls at home in patients with perineural femoral catheters: a retrospective summary of a randomized clinical trial. Anesth Analg. 2007 Apr;104(4):1002. doi: 10.1213/01.ane.0000256006.46703.7f. No abstract available. PMID 17377133
- [Background] Church S, Robinson TN, Angles EM, Tran ZV, Wallace JI. Postoperative falls in the acute hospital setting: characteristics, risk factors, and outcomes in males. Am J Surg. 2011 Feb;201(2):197-202. doi: 10.1016/j.amjsurg.2009.12.013. Epub 2010 Sep 18. PMID 20851375
- [Background] Lund J, Jenstrup MT, Jaeger P, Sorensen AM, Dahl JB. Continuous adductor-canal-blockade for adjuvant post-operative analgesia after major knee surgery: preliminary results. Acta Anaesthesiol Scand. 2011 Jan;55(1):14-9. doi: 10.1111/j.1399-6576.2010.02333.x. Epub 2010 Oct 29. PMID 21039357
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Background] Kennedy JC, Alexander IJ, Hayes KC. Nerve supply of the human knee and its functional importance. Am J Sports Med. 1982 Nov-Dec;10(6):329-35. doi: 10.1177/036354658201000601. PMID 6897495
- [Background] Franco CD, Buvanendran A, Petersohn JD, Menzies RD, Menzies LP. Innervation of the Anterior Capsule of the Human Knee: Implications for Radiofrequency Ablation. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):363-8. doi: 10.1097/AAP.0000000000000269. PMID 26066383
- [Background] Krenzel BA, Cook C, Martin GN, Vail TP, Attarian DE, Bolognesi MP. Posterior capsular injections of ropivacaine during total knee arthroplasty: a randomized, double-blind, placebo-controlled study. J Arthroplasty. 2009 Sep;24(6 Suppl):138-43. doi: 10.1016/j.arth.2009.03.014. Epub 2009 Jun 10. PMID 19520544
- [Background] C. Vlessides M. New Regional Technique Controls Post-TKA Pain. Anesthesiology News. December 2012.
- [Background] Egeler C, Jayakumar A, Ford S. Motor-sparing knee block - description of a new technique. Anaesthesia. 2013 May;68(5):542-3. doi: 10.1111/anae.12233. No abstract available. PMID 23573861
- [Background] Mantripragada S. A lipid based depot (DepoFoam technology) for sustained release drug delivery. Prog Lipid Res. 2002 Sep;41(5):392-406. doi: 10.1016/s0163-7827(02)00004-8. PMID 12121719
- [Background] Richard BM, Newton P, Ott LR, Haan D, Brubaker AN, Cole PI, Ross PE, Rebelatto MC, Nelson KG. The Safety of EXPAREL (R) (Bupivacaine Liposome Injectable Suspension) Administered by Peripheral Nerve Block in Rabbits and Dogs. J Drug Deliv. 2012;2012:962101. doi: 10.1155/2012/962101. Epub 2012 Jan 17. PMID 22363842
- [Background] Golf M, Daniels SE, Onel E. A phase 3, randomized, placebo-controlled trial of DepoFoam(R) bupivacaine (extended-release bupivacaine local analgesic) in bunionectomy. Adv Ther. 2011 Sep;28(9):776-88. doi: 10.1007/s12325-011-0052-y. Epub 2011 Aug 12. PMID 21842428
- [Background] Haas E, Onel E, Miller H, Ragupathi M, White PF. A double-blind, randomized, active-controlled study for post-hemorrhoidectomy pain management with liposome bupivacaine, a novel local analgesic formulation. Am Surg. 2012 May;78(5):574-81. doi: 10.1177/000313481207800540. PMID 22546131
- [Background] Gorfine SR, Onel E, Patou G, Krivokapic ZV. Bupivacaine extended-release liposome injection for prolonged postsurgical analgesia in patients undergoing hemorrhoidectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2011 Dec;54(12):1552-9. doi: 10.1097/DCR.0b013e318232d4c1. PMID 22067185
- [Background] Bergese SD, Ramamoorthy S, Patou G, Bramlett K, Gorfine SR, Candiotti KA. Efficacy profile of liposome bupivacaine, a novel formulation of bupivacaine for postsurgical analgesia. J Pain Res. 2012;5:107-16. doi: 10.2147/JPR.S30861. Epub 2012 May 1. PMID 22570563
- [Background] Ilfeld BM, Viscusi ER, Hadzic A, Minkowitz HS, Morren MD, Lookabaugh J, Joshi GP. Safety and Side Effect Profile of Liposome Bupivacaine (Exparel) in Peripheral Nerve Blocks. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):572-82. doi: 10.1097/AAP.0000000000000283. PMID 26204387
- [Background] Emerson RH Jr, Barrington JW, Olugbode O, Lovald S, Watson H, Ong K. Femoral Nerve Block Versus Long-Acting Wound Infiltration in Total Knee Arthroplasty. Orthopedics. 2016 May 1;39(3):e449-55. doi: 10.3928/01477447-20160315-03. Epub 2016 Mar 29. PMID 27018607
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Haley SM, Coster WJ, Andres PL, Ludlow LH, Ni P, Bond TL, Sinclair SJ, Jette AM. Activity outcome measurement for postacute care. Med Care. 2004 Jan;42(1 Suppl):I49-61. doi: 10.1097/01.mlr.0000103520.43902.6c. PMID 14707755
- [Background] Jette DU, Stilphen M, Ranganathan VK, Passek SD, Frost FS, Jette AM. AM-PAC "6-Clicks" functional assessment scores predict acute care hospital discharge destination. Phys Ther. 2014 Sep;94(9):1252-61. doi: 10.2522/ptj.20130359. Epub 2014 Apr 24. PMID 24764073
- [Background] Menendez ME, Schumacher CS, Ring D, Freiberg AA, Rubash HE, Kwon YM. Does "6-Clicks" Day 1 Postoperative Mobility Score Predict Discharge Disposition After Total Hip and Knee Arthroplasties? J Arthroplasty. 2016 Sep;31(9):1916-20. doi: 10.1016/j.arth.2016.02.017. Epub 2016 Feb 17. PMID 26993155
- [Background] Bickler P, Brandes J, Lee M, Bozic K, Chesbro B, Claassen J. Bleeding complications from femoral and sciatic nerve catheters in patients receiving low molecular weight heparin. Anesth Analg. 2006 Oct;103(4):1036-7. doi: 10.1213/01.ane.0000237230.40246.44. PMID 17000826
- [Background] Buckenmaier CC 3rd, Shields CH, Auton AA, Evans SL, Croll SM, Bleckner LL, Brown DS, Stojadinovic A. Continuous peripheral nerve block in combat casualties receiving low-molecular weight heparin. Br J Anaesth. 2006 Dec;97(6):874-7. doi: 10.1093/bja/ael269. Epub 2006 Oct 9. PMID 17032662
- [Background] Idestrup C, Sawhney M, Nix C, Kiss A. The incidence of hematoma formation in patients with continuous femoral catheters following total knee arthroplasty while receiving rivaroxaban as thromboprophylaxis: an observational study. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):414-7. doi: 10.1097/AAP.0000000000000127. PMID 25102065
- [Background] Brull R, McCartney CJ, Chan VW, El-Beheiry H. Neurological complications after regional anesthesia: contemporary estimates of risk. Anesth Analg. 2007 Apr;104(4):965-74. doi: 10.1213/01.ane.0000258740.17193.ec. PMID 17377115

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivicaine | Bupivicaine + Exparel
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivicaine | Bupivicaine + Exparel | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 6 | 6
  >=65 years | 13 | 6 | 19
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [66 to 75] | 67 [58 to 77] | 70 [63 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: AM-PAC Score to Measure Patients Fitness for Discharge
Description: AM-PAC (activity measure for post-acute care) will be used to determine if a patient is fit to discharge based on mobility with 6 being unable to mobilize up to 24 being independent. Patients who scored above 20 were considered fit to discharge.
Time Frame: Post-Operation Day 1
Measure: Mean (Inter-Quartile Range); unit: score on scale
Arm/Group | Bupivicaine | Bupivicaine + Exparel
Number analyzed (Participants) | 13 | 12
score on scale | 23 [19 to 23] | 23 [21 to 24]

2. Secondary Outcome: Opioid Consumption During the First 48 Hours After TKA Surgery
Description: Monitor how much opioid patient consumes
Time Frame: During the first 48 hours after surgery
Measure: Mean (Inter-Quartile Range); unit: milligram
Arm/Group | Bupivicaine | Bupivicaine + Exparel
Number analyzed (Participants) | 13 | 12
milligram | 90 [39 to 118] | 76 [25 to 128]

3. Secondary Outcome: Pain Scores During 48 Hrs Postoperatively
Description: Will use Numeric Pain Rating Scale (NPRS) to measure pain with 0 being no pain and 10 being the worst pain.
Time Frame: 48 hours postoperatively
Measure: Mean (Inter-Quartile Range); unit: score on scale
Arm/Group | Bupivicaine | Bupivicaine + Exparel
Number analyzed (Participants) | 13 | 12
score on scale | 4 [2.5 to 7] | 4 [3 to 5]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up until 48 hours post operation.
Arm/Group | Bupivicaine | Bupivicaine + Exparel
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT03303794/Prot_SAP_000.pdf